CLINICAL TRIAL: NCT00045149
Title: Phase I Study to Evaluate the Safety of Cellular Adoptive Immunotherapy Using Autologous CD8+ Antigen Specific T Cell Clones Targeting Cancer Testis Antigens for Patients With Metastatic Melanoma
Brief Title: Biological Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1588.00; FHCRC-1588.00; NCI-H02-0091; CDR0000256451 (Registry Identifier: PDQ); NCT00029432 (obsolete NCT alias)
Record Dates: First submitted 2002-09-06; First posted 2003-05-28 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-05

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Biological: therapeutic tumor infiltrating lymphocytes

SUMMARY:
RATIONALE: Biological therapies such as cellular adoptive immunotherapy use different ways to stimulate the immune system and stop cancer cells from growing. Treating a person's white blood cells in the laboratory and then reinfusing them may cause a stronger immune response and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of biological therapy in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and toxicity of cellular adoptive immunotherapy comprising autologous CD8+ cytotoxic T-lymphocyte clones targeting cancer-testis antigens in patients with metastatic melanoma.
* Determine the duration of in vivo persistence of this therapy in these patients.

Secondary

* Evaluate the antitumor effects of this therapy in these patients.

OUTLINE: Patients undergo leukapheresis to obtain peripheral blood mononuclear cells and then CD8+ cytotoxic T-lymphocyte (CTL) clones are generated ex vivo. Patients receive cellular adoptive immunotherapy comprising autologous CD8+ CTL clones targeting cancer testis antigens IV over 30 minutes on day 1. Patients also receive interleukin-2 subcutaneously every 12 hours on days 1-14 of courses 2-4. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients who demonstrate a clinical response after completion of the fourth course are eligible to receive additional T-cell infusions.

Patients are followed for 9 months.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma

  * Stage IV disease
* HLA-A1, -A2, and -A3 positive
* MAGE-1 or -3 positive by histology
* Bidimensionally measurable disease by palpation on clinical examination, x-ray, or CT scan
* No CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* Karnofsky 80-100%

Life expectancy

* More than 6 months

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 1.6 mg/dL
* SGOT ≤ 3 times upper limit of normal
* PT ≤ 1.5 times control

Renal

* Creatinine ≤ 2.0 mg/dL
* Calcium ≤ 12 mg/dL

Cardiovascular

* No congestive heart failure
* No clinically significant hypotension
* No symptoms of coronary artery disease
* No cardiac arrhythmias on electrocardiogram requiring drug therapy
* Patients with prior cardiovascular disease or the presence of any of the above abnormalities undergo a cardiac evaluation, which may include a stress test and/or echocardiogram

Pulmonary

* No clinically significant pulmonary dysfunction by medical history or physical examination
* FEV_1 ≥ 60% of normal
* DLCO ≥ 55% (corrected for hemoglobin)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No retinitis or choroiditis
* No active infections or oral temperature greater than 38.2 degrees Celsius within the past 72 hours
* No systemic infection requiring chronic maintenance or suppressive therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent immunotherapy (e.g., other interleukins, interferons, melanoma vaccines, intravenous immunoglobulin, or expanded polyclonal tumor-infiltrating lymphocytes or lymphokine-activated killer cell therapy)

Chemotherapy

* At least 3 weeks since prior standard or experimental chemotherapy
* 1-2 courses of prior cytoreductive chemotherapy for bulky disease allowed

Endocrine therapy

* No concurrent systemic steroids (except for toxicity management)

Radiotherapy

* At least 3 weeks since prior radiotherapy

Surgery

* Not specified

Other

* At least 3 weeks since prior immunosuppressive therapy
* No concurrent pentoxifylline
* No other concurrent investigational agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cassian Yee, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States